CLINICAL TRIAL: NCT02506686
Title: Evaluation of Meropenem Penetration Across Blood-Brain Barrier in Patients With Central Nervous System Infection After Neurosurgery and Optimization of Meropenem Treatment
Brief Title: Meropenem Penetration Across BBB in Patients With CNS Infection and Optimization of Meropenem Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jufang Wu, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MERO0001
Record Dates: First submitted 2015-07-17; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Central Nervous System Infections
MeSH Terms: conditions — Central Nervous System Infections | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Meropenem (Experimental): Meropenem i.v.
  Interventions: Drug: Meropenem

INTERVENTIONS:
Drug: Meropenem — Meropenem i.v.
  Other Names: Mero

SUMMARY:
A prospective, open-label study investigated the pharmacokinetic profile of meropenem in patients with post-neurosurgical central nervous system (CNS) infection, especially its BBB penetration into cerebrospinal fluid (CSF).

DETAILED DESCRIPTION:
Meropenem is important for management of post-neurosurgical meningitis, but the data about its penetration across blood-brain barrier (BBB) are inadequate. This prospective, open-label study investigated the pharmacokinetic profile of meropenem in patients with post-neurosurgical central nervous system (CNS) infection, especially its BBB penetration into cerebrospinal fluid (CSF). A total of 82 patients with post-neurosurgical CNS infection were included to receive meropenem intravenously according to regimen of 2g q8h, 1g q8h or 1g q6h. After infusion of 4 doses, blood and CSF samples were collected simultaneously at predefined timepoints. High-performance liquid chromatography ultraviolet method was used to determine the concentration of meropenem.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* requiring continuous drainage of CSF or gram-negative bacteria were identified from CSF culture
* have temperature fever (T > 37.5℃)
* have signs of meningeal irritation
* white blood cells in CSF > 300 × 10^6/L

Exclusion Criteria:

* hypersensitive to meropenem
* did not receive at least 3 days of meropenem treatment
* are receiving hemodialysis
* unstable vital signs
* have lumbar puncture contraindications and so inappropriate for sample collection
* severe hepatic or renal dysfunction
* status epilepticus
* potential neurodegenerative diseases
* pregnancy
* breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Concentrations of meropenem in plasma and CSF in patients with CNS Infections | Up to 12 months
  The concentrations of meropenem in plasma and CSF in patients with post-neurosurgical CNS after administration of three different dosing regimens of meropenem at each time points by HPLC-UV

CONTACTS AND LOCATIONS:
Overall Officials: Jufang Wu, MD, Principal Investigator — Huashan Hospital

REFERENCES:
- [Derived] Lu C, Zhang Y, Chen M, Zhong P, Chen Y, Yu J, Wu X, Wu J, Zhang J. Population Pharmacokinetics and Dosing Regimen Optimization of Meropenem in Cerebrospinal Fluid and Plasma in Patients with Meningitis after Neurosurgery. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6619-6625. doi: 10.1128/AAC.00997-16. Print 2016 Nov. PMID 27572392